CLINICAL TRIAL: NCT06869655
Title: Resistive Diaphragmatic Training Versus Volumes Oriented Spirometry On Pulmonary Function Test And Functional Capacity In Asthmatic Patients.
Brief Title: Resistive Diaphragmatic Training vs Volumes-Oriented Spirometer In Asthmatic Parients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0321 Maria
Record Dates: First submitted 2025-02-20; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: Diaphragm training; Pulmonary function test; Rehabilitation; Spirometry; Six-minute walk test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Threshold Loading device (Experimental): Resistive Diaphragmatic Training: In this group of participants will receive resistive diaphragm training with the help of threshold loading device along conventional physiotherapy under supervision for 6 weeks.
  Interventions: Device: Threshold Loading device
- Volumes Oriented Spirometry (Experimental): volume-oriented incentive spirometry: In this group of participants will receive training through volume-oriented incentive spirometer emphasizing lung capacity and airflow along with conventional physiotherapy under supervision for 6 weeks.
  Interventions: Device: Volumes Oriented Spirometry

INTERVENTIONS:
Device: Threshold Loading device — threshold loading device for diaphragmatic resistance training
  Arms: Threshold Loading device
Device: Volumes Oriented Spirometry — group B will receive this interentions
  Arms: Volumes Oriented Spirometry

SUMMARY:
Asthma, a chronic lung disease characterized by airway inflammation and constriction, presents ongoing challenges despite advancements in treatment. The aim of this study to deliver non-pharmacological interventions, particularly comparing resistive diaphragmatic training (RDT) and volume-oriented spirometry, to assess their efficacy in enhancing pulmonary function and functional capacity among asthmatic patients. it will compare resistive diaphragmatic training (RDT) with volume-oriented spirometry in asthmatic patients to pinpoint the superior method for enhancing lung function and daily capabilities.

DETAILED DESCRIPTION:
Asthma is a chronic lung disease characterized by airway inflammation and constriction, presents ongoing challenges despite advancements in treatment.The aim of this study is to deliver non-pharmacological interventions, comparing resistive diaphragmatic training (RDT) and volume-oriented spirometry, to assess their efficacy in enhancing pulmonary function and functional capacity among asthmatic patients. Method: This study will be conducted at "Gulab Devi Chest Hospital" Lahore, it is randomized clinical trial (RCT) which will divided into two groups: Group A include RDT along conventional physiotherapy treatment and Group B include volume-oriented spirometry along conventional physiotherapy treatment. Total 50 subjects will be recruited according inclusion and exclusions criteria by convenient sampling technique. Data collection procedure will follow standardized procedures like pre-assessment and post-assessment which will be after 6 weeks with spirometry, 6MWT, and the ACT. Hypothesis postulated that RDT will show greater mprovements in pulmonary function and functional capacity compared to volumes oriented spirometry. However, null hypothesis will suggest that there is no significant difference between the two interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 35 years to 50 years who must have a confirm diagnosis of asthma and FEV1% >60% & <80%, both male and female with moderate asthma. Outpatients from regional medical Centre.

Exclusion Criteria:

* Asthma patients whose condition require hospitalization asthmatic patients with physical limitation patients, with exercise-induced asthma, Asthma patients with heart dis¬ease with evidence of cardiovascular osteoarticular, inability to consent or cooperate, long-term, home oxygen therapy, active tuberculosis or other infectious disorders as well as stroke, are excluded

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
6-MWT | 6-weeks
  For the 6MWT assessment, the participants were encouraged to walk as far as they could during 6 min over a flat 100-feet surface, and for consistency, the researchers used constant verbal cues and positive feedback to encourage the participants to complete the task. The 6-Minute Walk Test (6MWT) assesses aerobic capacity and functional exercise capacity by measuring the distance a person can walk in 6 minutes. Results are interpreted based on the distance walked, which correlates with functional capacity.
Asthma Control Test | 6-weeks
  The ACT is a validated, patient-completed measure of asthma control that includes five questions that assess activity limitations, shortness of breath, nighttime symptoms, use of rescue medication, and patient overall rating of asthma control over the previous four weeks. The questions are scored from 1 (worst) to 5 (best), and the ACT score is the sum of the responses, giving a maximum best score of 25.
spirometer | 6-weeks
  For Pulmonary Function, FEV1 will be used to assess lung function. A spirometer will be used to measure forced expiratory volume in 1 second (FEV1). The spirometer is a simple test and an essential tool in diagnosing airway obstruction. However, the variability of spirometry measurements is greater than in most other clinical laboratory tests because the result is highly dependent on the consistency of the efforts made by patients and technicians. Normal values vary based on age, sex, height, and ethnicity. Interpretations are based on comparing results to predicted values, aiding in diagnosing conditions like asthma or COPD. However, interpretation accuracy can also depend on the expertise of the interpreter and clinical context. For instance: FVC: Around 80-120% of predicted value, FEV1: Around 75-85% of predicted value and FEV1/FVC ratio: Typically >0.7 (adults).

CONTACTS AND LOCATIONS:
Overall Officials: Qurat Ul Ain, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Lima FF, Pinheiro DHA, de Carvalho CRF. Physical training in adults with asthma: An integrative approach on strategies, mechanisms, and benefits. Front Rehabil Sci. 2023 Feb 17;4:1115352. doi: 10.3389/fresc.2023.1115352. eCollection 2023. PMID 36873818
- [Background] Aegerter H, Lambrecht BN. The Pathology of Asthma: What Is Obstructing Our View? Annu Rev Pathol. 2023 Jan 24;18:387-409. doi: 10.1146/annurev-pathol-042220-015902. Epub 2022 Oct 21. PMID 36270294
- [Background] Mosnaim G. Asthma in Adults. N Engl J Med. 2023 Sep 14;389(11):1023-1031. doi: 10.1056/NEJMcp2304871. No abstract available. PMID 37703556
- [Background] Ramos E, de Oliveira LV, Silva AB, Costa IP, Correa JC, Costa D, Alves VL, Donner CF, Stirbulov R, Arena R, Sampaio LM. Peripheral muscle strength and functional capacity in patients with moderate to severe asthma. Multidiscip Respir Med. 2015 Jan 21;10(1):3. doi: 10.1186/2049-6958-10-3. eCollection 2015. PMID 25973197
- [Background] Chung Y, Huang TY, Liao YH, Kuo YC. 12-Week Inspiratory Muscle Training Improves Respiratory Muscle Strength in Adult Patients with Stable Asthma: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Mar 22;18(6):3267. doi: 10.3390/ijerph18063267. PMID 33809922